CLINICAL TRIAL: NCT02102529
Title: Survey: Clinical Outcome After Bowel Resection in Women Due to Endometriosis
Status: Completed | Type: Observational
Sponsor: Kepler University Hospital (Other)
Responsible Party: Principal Investigator, Klugsberger Bettina, M.D., Ludwig Boltzmann Institute for Operative Laparoscopy
Other Study IDs: ENCO-014; ENCO-014 (Other: 2nd Surgical Department, General Hospital, Linz)
Record Dates: First submitted 2014-03-30; First posted 2014-04-03 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Bowel Endometriosis
Keywords: pain; quality of life
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- bowel endometriosis: laparoscopic colonic resection
  Interventions: Procedure: laparoscopic colonic surgery

INTERVENTIONS:
Procedure: laparoscopic colonic surgery — women with typical symptoms including pelvic pain, infertility and endometriotic bowel lesions who underwent laparoscopic surgery including colonic resection performed from 2009 to 2012

SUMMARY:
Endometriosis is one of the most frequent benign diseases that can affect women in their reproductive age. In severe form, the colon or rectum may be involved. It has been shown that the surgical treatment improve typical symptoms like pain and dyspareunia. The investigators evaluated the functional results and quality of life after laparoscopic colonic resection for endometriosis

DETAILED DESCRIPTION:
A clinical analysis of thirty women with typical symptoms including pelvic pain, infertility and endometriotic bowel lesions who underwent laparoscopic surgery including colonic resection performed from 2009 to 2012. Quality of life and pain was documented postoperatively. We conduct a telephone survey, which starts at May 2014.

ELIGIBILITY:
Inclusion Criteria:

* •Clinical diagnosis of endometriosis

Exclusion Criteria:

* Unwillingness to participate on the survey

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women with typical symptoms including pelvic pain, infertility and endometriotic bowel lesions who underwent laparoscopic surgery including colonic resection performed from 2009 to 2012
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-04; Primary Completion 2016-08 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
visual analog scala for pain | one year after the operation
  comparison of pain before and after the operation (one year later), value 0 til 10; 0= no pain, 10= strong pain

SECONDARY OUTCOMES:
dyspareunia | one year after the operation
  comparison of dyspareunia before and one year after the operation
dysuria | one year after operation
  comparison of dysuria before and one year after the operation
obstipation | one year after operation
  comparison of obstipation before and one year after the operation
pain during defecation | one year after operation
  comparison of pain during defecation before and one year after the operation
rectal bleeding | one year after operation
  comparison of rectal bleeding during menstruation before and one year after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Shamiyeh, Univ-Prof.Dr, Study Chair — Ludwig Boltzmann Institute for Operative Laparoscopy, 2nd Surgical Department, Academic Teaching Hospital, AKH Linz
Locations (1):
- 2nd Surgical Department, Academic Teaching Hospital, AKH Linz, Linz, Upper Austria, Austria

REFERENCES:
- [Result] Haas D, Chvatal R, Habelsberger A, Wurm P, Schimetta W, Oppelt P. Comparison of revised American Fertility Society and ENZIAN staging: a critical evaluation of classifications of endometriosis on the basis of our patient population. Fertil Steril. 2011 Apr;95(5):1574-8. doi: 10.1016/j.fertnstert.2011.01.135. PMID 21315335